CLINICAL TRIAL: NCT07075068
Title: The Effects of Cigarette Addiction on Lower Extremity Movement Speed and Coordination in Young Adults
Brief Title: The Effects of Cigarette Addiction on Lower Extremity Movement Speed and Coordination
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: Smoking&Speed
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smokers: Individuals who will meet WHO and DSM-IV-TR criteria for cigarette dependence.
  Interventions: Diagnostic Test: Behavioral and Functional Performance Assessment Battery
- Non-Smokers: Individuals who will report no smoking behavior in the past year.
  Interventions: Diagnostic Test: Behavioral and Functional Performance Assessment Battery

INTERVENTIONS:
Diagnostic Test: Behavioral and Functional Performance Assessment Battery — This study will include only observational functional assessments. No active intervention will be performed.This observational protocol will involve standardized assessments of lower extremity coordination (LEMOCOT), movement speed (30-meter sprint), and smoking-related behavioral patterns (Fagerström Test for Nicotine Dependence). These tools will be used to evaluate the potential impact of cigarette addiction on physical performance in young adults. No therapeutic or pharmacological intervention will be applied.

SUMMARY:
This observational study will aim to investigate the effects of cigarette addiction on lower extremity motor coordination and movement speed in young adults. The study will include healthy participants aged 18-25 years, divided into smokers and non-smokers. Motor coordination will be assessed using the Lower Extremity Motor Coordination Test (LEMOCOT), and speed will be evaluated with a 30-meter sprint test. Nicotine dependence will be evaluated in smokers using the Fagerström Test. The findings will provide insight into the possible functional impacts of nicotine addiction on motor performance.

DETAILED DESCRIPTION:
The study will be conducted as a non-randomized controlled observational trial at the Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation. A total of 24 healthy young adults (12 smokers, 12 non-smokers) will participate. The inclusion criteria will require participants to be aged 18-25, cooperative, literate, and able to walk independently. Participants will be categorized as smokers based on WHO and DSM-IV-TR criteria. The primary assessments will include LEMOCOT and 30-meter sprint test. Nicotine addiction will be measured using the Fagerström Test for Nicotine Dependence (FTND), and anthropometric data including BMI and bimalleolar diameter will also be recorded. Data will be analyzed to determine any statistical differences or correlations between smoking status and motor performance outcomes.

ELIGIBILITY:
Inclusion Criteria (for both groups):

* Age between 18 and 25 years
* Able to walk independently
* Literate and cooperative
* Willing to participate voluntarily
* BMI between 18.5 and 29.9 kg/m²

Additional inclusion for smokers:

* Daily smoking for at least one year based on WHO and DSM-IV-TR definitions
* Exclusion Criteria (for all participants):
* Orthopedic, neurologic, or neuromuscular disorders affecting gait
* Chronic cardiopulmonary disease
* Cognitive impairments
* Obesity (BMI ≥ 30 kg/m²)

Additional exclusion for smokers:

* History of acute cardiovascular events
* Chronic heart failure or lung diseases

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: The study population will consist of healthy young adults aged between 18 and 25 years. A total of 24 participants will be included, with 12 individuals who meet the criteria for cigarette dependence and 12 who do not smoke. Participants will be recruited from a university setting using convenience and snowball sampling methods. All participants will be required to be cooperative, literate, and able to walk independently. They will also be screened to ensure a body mass index (BMI) between 18.5 and 29.9 kg/m². Smokers will be identified based on the World Health Organization (WHO) definition and the DSM-IV-TR diagnostic criteria. Individuals with orthopedic, neurologic, cardiopulmonary, or cognitive impairments will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
LEMOCOT Score (Lower Extremity Motor Coordination Test) | Baseline
  The number of correct taps within 20 seconds will be measured for each participant.
30-Meter Sprint Time | Baseline
  Time (in seconds) required to complete a 30-meter sprint will be recorded and averaged from two trials.

SECONDARY OUTCOMES:
Fagerström Test for Nicotine Dependence Score | Baseline
  Degree of nicotine dependence will be evaluated in smokers using the Fagerström Test for Nicotine Dependence.
Body Mass Index (BMI) | Baseline
  BMI will be calculated using height and weight measurements (BMI = weight (kg) / height² (m²)).
Bimalleolar Circumference and Diameter Measurement | Baseline
  The circumference at the level of the medial and lateral malleoli will be measured using a flexible tape measure while the participant is in a supine position.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehlivan, Istanbul, Üsküdar, Turkey (Türkiye)